CLINICAL TRIAL: NCT05453682
Title: Hypofractionated Intensity-modulated Radiation Therapy With Concurrent Chemotherapy in Musc Le-invasive Bladder Cancer:
Brief Title: Hypofractionated IMRT With Concurrent Chemotherapy in Muscle-invasive Bladder Cancer (HIRACUM)
Acronym: HIRACOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Park, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC-2021-01-026
Record Dates: First submitted 2021-12-29; First posted 2022-07-12 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; hypofractionated radiotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypo IMRT (Experimental): in muscle invasive bladder cancer, hypofractionated IMRT with chemotherapy
  Interventions: Radiation: hypo-IMRT

INTERVENTIONS:
Radiation: hypo-IMRT — Twenty fractionation within 4 weeks are performed using hypofractionated intensity-modulated radiation therapy. As for the radiation dose, 2.8-3.2 Gy at a time, total dose 56-64 Gy, to the high-risk target volume, and 2-2.2 Gy at a time, and 40-44 Gy, respectively, to the low-risk target volume.

SUMMARY:
The purpose of this study is to investigate the side effects, quality of life, and treatment effects of concurrent chemo-hypofractionated intensity-modulated radiation therapy in bladder cancer.

Twenty fractionation within 4 weeks are performed using hypofractionated intensity-modulated radiation therapy. As for the radiation dose, 2.8-3.2 Gy at a time, total dose 56-64 Gy, to the high-risk target volume, and 2-2.2 Gy at a time, and 40-44 Gy, respectively, to the low-risk target volume. It aims to include more than 97% of the total dose to cover the entire PTV, and the minimum dose in the PTV is not lower than 95% of the prescribed dose, and the maximum dose does not exceed 107% of the prescribed dose. Chemotherapy before and after radiotherapy can be performed depending on the institutional policy. Among radiotherapy, chemotherapy is performed with platinum-based agents (cisplatin, carboplatin, etc.), and is administered once a week for a total of 3 or more.

DETAILED DESCRIPTION:
For bladder cancer, conventional concurrent chemoradiotherapy is irradiated with a daily radiation dose of 1.8-2.0 Gy each, a total of 64 Gy or more, and the radiation treatment period takes more than 6 weeks in bladder preserving protocol. Concurrent chemoradiotherapy has the advantage of bladder preservation, but gastrointestinal, genitourinary, and hematologic side effects occur in about 5%. Hypofractionated radiotherapy has the advantage of increasing the radiation-biological effect on tumors by reducing the number of treatments instead of increasing the daily dose, and shortening the overall treatment time. On the other hand, hypofractionated radiotherapy can also increase the risk of side effects related to treatment because the radiologic effects on normal tissues also increase. However, the biological effect of radiation on normal tissues can be reduced by applying intensity-modulated radiation therapy in hypofractional radiation therapy to reduce radiation exposure to normal tissues. Clinical studies of concurrent chemotherapy with hypofractionation radiation therapy are still in its insignificant stage.

The purpose of this study is to investigate the side effects, quality of life, and treatment effects of concurrent chemo-hypofractionated intensity-modulated radiation therapy in bladder cancer.

The 2-year bladder conserving disease-free survival rate after the existing concurrent chemo-radiation therapy is known to be about 55%, and when concurrent chemo-hyofractionated intensity-modulated radiation therapy is performed in invasive bladder cancer, the 2-year bladder conservation disease-free survival rate is expected about 70%. The number of patients required to verify this was 80% power, a significance level of alpha = 0.1, recruitment of patients for 3 years, and taking into account the follow-up observation for 2 years after recruitment, and setting the dropout rate of 15%, a total of 53 patients was necessary.

Twenty fractionation within 4 weeks are performed using hypofractionated intensity-modulated radiation therapy. As for the radiation dose, 2.8-3.2 Gy at a time, total dose 56-64 Gy, to the high-risk target volume, and 2-2.2 Gy at a time, and 40-44 Gy, respectively, to the low-risk target volume. It aims to include more than 97% of the total dose to cover the entire PTV, and the minimum dose in the PTV is not lower than 95% of the prescribed dose, and the maximum dose does not exceed 107% of the prescribed dose. Chemotherapy before and after radiotherapy can be performed depending on the institutional policy. Among radiotherapy, chemotherapy is performed with platinum-based agents (cisplatin, carboplatin, etc.), and is administered once a week for a total of 3 or more.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with bladder cancer histologically
2. Patients with muscle layer involvement in transurethral resection (pT2 or higher)
3. Patients without pelvic lymph node metastasis by computed tomography (CT) or magnetic resonance images (MRI) of the pelvis.
4. Patients who want bladder conservation treatment
5. Patients over 20 years old
6. Patients with Zubrod (ECOG) performance status 0-1 within 1 week prior to participation in the study
7. Patients who have signed the consent form with sufficient information by the patient or guardian
8. Patients with hematologic findings capable of concurrent chemoradiotherapy

Exclusion Criteria:

1. Patients with previous pelvic radiotherapy history
2. Pregnant or lactating patients
3. Patients with distant metastasis
4. Patients judged to be difficult to conserve bladder due to extensive non-invasive/invasive bladder cancer
5. Patients who have not been disease-free for more than 5 years after diagnosis of cancer (excluding thyroid cancer, non-melanoma skin cancer, T1a prostate cancer, and intraepithelial cancer of the cervix)
6. Patients with untreated severe acute disease
7. Patients predicted to have a high probability of radiation complications due to connective tissue disease (lupus, scleroderma, etc.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
bladder preservation disease-free survival rate | 2 years after participation of all subjects
  Two-year bladder preservation disease-free survival rate when concurrent chemo-hypofractionated intensity-modulated radiation therapy

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Number of participants with treatment-related adverse events as assessed CTCAE v5.0 radiation therapy | 3 months after participation
  acute toxicity
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0radiation therapy | 5 years after participation
  late toxicity
EORTC QOL-C30 measurement | 5 years after participation
  QoL
2 year disease-free survival when concurrent chemo-hypofractionated intensity-modulated radiation therapy | 2 years after participation of all subjects
  disease-free survival
overall survival when concurrent chemo-hypofractionated intensity-modulated radiation therapy | 5 years after participation of all subjects
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided